CLINICAL TRIAL: NCT01961245
Title: Effects of Nocturnal Non-invasive Ventilation on Energy Expenditure in Patients With Severe Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Dr., Schön Klinik Berchtesgadener Land
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BGL-NIV2
Record Dates: First submitted 2013-09-30; First posted 2013-10-11 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Rehabilitation; Non-invasive Ventilation; Energy Expenditure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- nocturnal non-invasive ventilation (Active Comparator): patients will undergo 12 nights of non-invasive ventilation during pulmonary rehabilitation
  Interventions: Device: nocturnal non-invasive ventilation
- no nocturnal non-invasive ventilation (No Intervention): patients will undergo pulmonary rehabilitation without nocturnal non-invasive ventilation

INTERVENTIONS:
Device: nocturnal non-invasive ventilation — patients will undergo a non-invasive ventilation during the night
  Arms: nocturnal non-invasive ventilation

SUMMARY:
It has been shown, that in patients with very severe chronic obstructive pulmonary disease (COPD) the additional use of non-invasive ventilation during pulmonary rehabilitation (PR) may enhance the benefits of PR. It is assumed that the non-invasive ventilation techniques provides a better recovery of the respiratory pump during the night. If non-invasive ventilation also decreases the metabolic demands during night is unknown and is aim of this study. During a 3 week inpatient pulmonary rehabilitation program a total of 85 patients with chronic obstructive pulmonary disease stage IV will be recruited for this study. There will be a 4:1 distribution into 2 groups. 68 patients with an indication for the use of a non-invasive ventilation will be involved in the intervention group where non-invasive ventilation will be initialized. 17 patients with chronic obstructive pulmonary disease stage IV without an indication for the use of non-invasive ventilation will be involved in a control group to detect the changes in nocturnal energy expenditure produced by pulmonary rehabilitation alone. All outcome measurements will be performed during day 1-3 and will be repeated after 12 days (with or without non-invasive ventilation) at day 15-17 of the pulmonary rehabilitation program.

A sub-trial of this study is to validate night movement accuracy of the Dynaport activity monitor with the observations made by a night-vision camera in the sleep lab. This will be performed in study participants as well as in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria for Intervention group:

* chronic obstructive pulmonary disease stage IV
* indication for the use of a nocturnal non-invasive ventilation (according to the German guidelines Schoenhofer et al. 2008)
* patient has not yet used non-invasive ventilation at all or inadequately (less than 3 hours per day)

Exclusion Criteria for Intervention group:

* acute exacerbation of chronic obstructive pulmonary disease
* severe heart failure
* body-mass-index >35 m²/kg
* fever

Inclusion Criteria for control group:

* chronic obstructive pulmonary disease stage IV (- healthy volunteers are also eligible for the sub-trial of this study to validate night movement accuracy of an activity monitor)

Exclusion Criteria for control group:

* acute exacerbation of chronic obstructive pulmonary disease
* indication for the use of a non-invasive ventilation
* severe heart failure
* body-mass-index >35 m²/kg
* fever

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2013-12 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
energy expenditure during night | day 1-3 and day 14-16
  energy expenditure will be assessed by Sensewear Armband

SECONDARY OUTCOMES:
energy expenditure during day | day 1-3 and day 14-16
  energy expenditure will be assessed by SenseWear Armband
lung function | day 1-3 and day 14-16
  measured by a bodyplethysmograph
sleep quality | day 1-3 and day 14-16
  measured by Severe Respiratory Insufficiency Questionnaire
arterial pressure of carbon dioxide during night | day 1-3 and day 14-16
  measured transcutaneously by a Sentec device
movement activity during the night | day 1
  night movement activity will be measured in a subgroup with the Dynaport device

CONTACTS AND LOCATIONS:
Locations (1):
- Schoen Klinik Berchtesgadener Land, Schönau am Königssee, Bavaria, Germany